CLINICAL TRIAL: NCT04689295
Title: The Effect of Schroth Method on Pain, Body Awareness and Quality of Life in Adolescent Individuals With Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Fatih Çelik, principal investigator, Hacettepe University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2019/0041
Record Dates: First submitted 2020-12-02; First posted 2020-12-30 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Scoliosis
Keywords: Schroth; idiopathic scoliosis; pain; quality of life; body awareness
MeSH Terms: conditions — Scoliosis; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experiment group (Other): Three dimensional scoliosis therapy method (Schroth) will be applied to the participants for 6 weeks. It consist of 15 different exercises combined with rotational breathing exercise.
  Interventions: Other: exercise programme 1
- control group (Other): Traditional scoliosis exercises will be applied to the participants for 6 weeks. It consist of 6 different exercises
  Interventions: Other: exercise programme 2

INTERVENTIONS:
Other: exercise programme 1 — Schroth three dimensional scoliosis therapy method
  Arms: experiment group
Other: exercise programme 2 — Traditional scoliosis exercises
  Arms: control group

SUMMARY:
This study was aimed to compare the effect of Schroth therapy method, which is a 3-dimensional scoliosis exercise method, and traditional exercises on pain, body awareness and quality of life in young individuals with idiopathic scoliosis.

DETAILED DESCRIPTION:
38 individuals aged between 10-18 with the diagnosis of idiopathic scoliosis will be participated in the study. Individuals (study group) underwent 1 hour exercise program 3 times a week for 6 weeks, and the individuals (control group) undervent a traditional exercise program once a week under supervision of physiotherapist for 6 weeks. During the rest of the week, same exercise program was given as a home program for at least half an hour a day and individuals will followed up. Individuals' subjective pain intensity will be assessed with Visual Analogue Scale (VAS), pressure pain threshold by algometer, body awareness by Turkish version of Body Awareness Questionnaire and quality of life by Turkish version of Scoliosis Research Society (SRS)-22 scale. Measurements will be performed before and after the 6-week exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with idiopathic scoliosis by a specialist physician,
* Between the ages of 10-18,
* Primary curvature between 20-40 degrees according to the Cobb method,
* Having C or S type of scoliosis,
* Having back / low-back pain due to scoliosis,
* Those who have not received any previous exercise therapy for scoliosis,
* Volunteering to participate in the study,
* Having the cognitive capacity to cooperate with the directions of the physiotherapist,
* Has not suffered any injuries to the musculoskeletal system in the last 6 months,
* No neurological, orthopedic or cardiopulmonary disorders other than scoliosis diagnosis,
* Young individuals who have not undergone any surgery related to the diagnosis of scoliosis

Exclusion Criteria:

* Previous spinal surgery,
* Any disease other than idiopathic scoliosis,
* Individuals who cannot adapt to the directions of the physiotherapist and cannot fulfill the requirements of the exercise program

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Pain Level | 6 weeks
  Pain level will be assessed with VAS (visual analog scale) (min:0, max:10)
Pressure Pain Threshold | 6 weeks
  Pressure pain threshold with algometer (kg/cm^2).

SECONDARY OUTCOMES:
Body awareness before and after treatment | 6 weeks
  body awareness assessment will be done with body awareness questionnaire (min:18, max:126 pts.)

OTHER OUTCOMES:
Quality of life before and after treatment | 6 weeks
  quality of life assessment will be done with SRS-22 (scoliosis research society 22 form)(min:1, max:5 pts.)

CONTACTS AND LOCATIONS:
Overall Officials: fatih çelik, Study Director — physiotherapist
Locations (1):
- Fizyo Omurga, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No